CLINICAL TRIAL: NCT07277673
Title: Is There a Benefit of Aerobic Exercise Addition to Cognitive Behavioural Treatment in Heavy Drinking Men With Impotence and Metabolic Syndrome?
Brief Title: Aerobic Exercise Addition to Cognitive Behavioural Treatment in Impotence Metabolic-syndrome Drinkers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB000-14233-55
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Heavy Drinking; Metabolic Syndrome; Impotence
MeSH Terms: conditions — Metabolic Syndrome; Erectile Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): Twenty men with Heavy Drinking, Impotence, and Metabolic Syndrome will be included. Men will receive Cognitive Behavioural Treatment (30 minute per the session , three times/week, for 12 weeks). Also, men will also adminsiter supervised aerobic training (walking on electrical treamill, 50 minute per the session, three times/week, for 12 weeks).
  Interventions: Behavioral: aerobci physical training and cognitive behavioural treatment
- group number 2 (Active Comparator): Twenty men with Heavy Drinking, Impotence, and Metabolic Syndrome will be included. Men will receive Cognitive Behavioural Treatment (30 minute per the session, three times/week, for 12 weeks).
  Interventions: Behavioral: Cognitive behavioural treatment

INTERVENTIONS:
Behavioral: aerobci physical training and cognitive behavioural treatment — Twenty men with Heavy Drinking, Impotence, and Metabolic Syndrome receive Cognitive Behavioural Treatment (30 minute per the session , three times/week, for 12 weeks). Also, men will also adminsiter supervised aerobic training (walking on electrical treamill, 50 minute per the session, three times/week, for 12 weeks).
  Arms: group number 1
Behavioral: Cognitive behavioural treatment — Twenty men with Heavy Drinking, Impotence, and Metabolic Syndrome will receive Cognitive Behavioural Treatment (30 minute per the session , three times/week, for 12 weeks)
  Arms: group number 2

SUMMARY:
Cognitive Behavioural Treatment is used as treatment for Heavy Drinking, Impotence, and Metabolic Syndrome. The efficacy of adding aerobic training to this treatment is not tested till now.

DETAILED DESCRIPTION:
Forty men with Heavy Drinking, Impotence, and Metabolic Syndrome will be included. catogorization will be performed to assign them to group number I or group number II. Every group will involve/contain twenty males. Both groups will receive Cognitive Behavioural Treatment (30 minute per the session , three times/week, for 12 weeks). Also, Group number I will also adminsiter supervised aerobic training (walking on electrical treamill, 50 minute per the session , three times/week, for 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* heavy drinking men (forty)
* men who complain metabolic syndrome
* men who complain impotence

Exclusion Criteria:

* cardiac problems
* renal or hepatic or respiratory or neurogenic diseases,

Ages: 35 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
international index of erectile function | it will be measured after 12 weeks
  it contain 5 questions that will assess penile erectile functions

SECONDARY OUTCOMES:
body mass index | It will be measured after 12 weeks
  it will be assessed on empty stomach and empty bladder and empty bowel
waist circumference | It will be measured after 12 weeks
  it will be assessed at ubmlilicus by a tape
blood systolic pressure | It will be measured after 12 weeks
  it will be assessed via sphygmonameter
blood diastolic pressure | it will be measured after 12 weeks
  it will be assessed via sphygmonameter
triglycerides | It will be measured after 12 weeks
  it will be assessed in plasma
high density lipoproteins | It will be measured after 12 weeks
  it will be assessed via plasma
blood glucose | It will be measured after 12 weeks
  it will assessed vin fasting plasma
Alcohol abstinence self-efficacy | It will be measured after 12 weeks
  the total score of this questionaire will be estimated
negative affect | It will be measured after 12 weeks
  a subscomponent of Alcohol-abstinence self-efficacy questioannire
Positive and social affect | It will be measured after 12 weeks
  a subscomponent of Alcohol-abstinence self-efficacy questioannire
physical and other concerns | It will be measured after 12 weeks
  a subscomponent of Alcohol-abstinence self-efficacy questioannire
craving and urges | It will be measured after 12 weeks
  a subscomponent of Alcohol-abstinence self-efficacy questioannire
Depression, Anxiety and Stress Scale | It will be measured after 12 weeks
  the total score of this questioannaire that contin 21 questions will be scored

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Dokki, Egypt